CLINICAL TRIAL: NCT06199323
Title: Acupuncture Therapy on Dysphagia in Parkinson's Disease: A Randomized Controlled Study
Brief Title: Acupuncture Therapy on Dysphagia in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-KS-HNSR008
Record Dates: First submitted 2023-12-20; First posted 2024-01-10 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All researchers were required to maintain isolation from participants beyond necessary contact and strictly keep confidentiality of research content. We used blind labels to identify participants' intervention or treatment allocation. These labels remained confidential during the research process and were accessible only to researchers and specific staff. In addition, all data collection and assessment were conducted by professionals who were not involved in the intervention and were not aware of the study design to ensure objectivity and independence. All medical staff responsible for the intervention received detailed training before the start of the study to ensure their understanding and proper implementation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment+swallowing rehabilitation training+acupuncture therapy (Experimental): The experimental group was given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given acupuncture therapy.
  Interventions: Behavioral: Routine rehabilitation training; Behavioral: Swallowing rehabilitation training; Procedure: Acupuncture therapy
- routine treatment+swallowing rehabilitation training (Active Comparator): The control group was given routine treatment and swallowing rehabilitation training.
  Interventions: Behavioral: Routine rehabilitation training; Behavioral: Swallowing rehabilitation training

INTERVENTIONS:
Behavioral: Routine rehabilitation training — 1. Balance function training: Patients were instructed to achieve weight shift between the left and right sides of the balance bar in a standing position.
  2. Walking function training: based on hip, knee, and ankle control training, patients were instructed to take steps training.
  3. Core muscle strength training: Patients were instructed to maintain 3 minutes of training in Bridge-style movement.
  4. Functional training of daily living: including training on dressing and undressing, independent eating, painting, and writing.
  Routine rehabilitation training was performed 30-45 minutes/time, 1-2 times/day, 5-7 days/week.
Behavioral: Swallowing rehabilitation training — 1. Swallowing-related organ training: including movement training of lip, mandibular muscle, cheek, tongue muscle, soft palate, as well as exercises of vocal cord closure, laryngeal lifting and pharyngeal muscle training. 5-15 minutes/time, 1-2 times/day, 5-7 days/week.
  2. Sensory stimulation training: With the self-made popsicle, medical staff slowly and gently stimulated the patient's cheek, palatoquadrate, soft palate, posterior pharyngeal wall, tongue surface and sublingual area repeatedly. 5-25 minutes/time, 1-3 times/day, 3-7 days/week.
  3. Direct training: When the patient's swallowing function improves to a certain extent of which the safety of oral intake can be basically ensured, oral feeding training (direct training) can be attempted gradually.
  4. Mendelsohn maneuver: During the Mendelsohn maneuver, the patient consciously prolonged the duration of the muscle contraction in the throat during swallowing.15-30 minutes/time, once per day, 5 days/week.
Procedure: Acupuncture therapy — The whole acupuncture therapy was performed once daily for 5 days per week, including acupuncture needle and tongue needle.
  Acupuncture needle:
  Main acupoints: Lianquan, Shanglianquan (depression between the hyoid bone and the lower border of the mandible), Yifeng; Auxiliary acupoints: Fengchi, Wangu, Fengfu, Yamen, Neidaying (depression of 1 inch below the anterior margin of the mandible).
  Tongue needle (pricking):
  Acupoints: Jinjin, Yuye, posterior pharyngeal wall (both sides of the uvula).
  Arms: routine treatment+swallowing rehabilitation training+acupuncture therapy

SUMMARY:
From June 2019 to May 2021, we conducted a randomized controlled study, including dysphagic patients with Parkinson's diseases who were admitted to the department of rehabilitation medicine in 3 hospitals in China. The participants were divided randomly into the experimental group and the control group, with 56 in each one. Both two groups were given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given acupuncture therapy.

DETAILED DESCRIPTION:
From June 2019 to May 2021, we conducted a randomized controlled study, including dysphagic patients with Parkinson's diseases who were admitted to the department of rehabilitation medicine in 3 hospitals in China. The participants were divided randomly into the experimental group and the control group, with 56 in each one. Both two groups were given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given acupuncture therapy. The study lasted 42 days (6 weeks) for each participant.

Specifically, our main focus is on the study of Lianquan, Shanglianquan (depression between the hyoid bone and the lower border of the mandible), Yifeng, Fengchi, Wangu, Fengfu, Yamen, Neidaying (depression of 1 inch below the anterior margin of the mandible), Jinjin, Yuye, posterior pharyngeal wall (both sides of the uvula).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the Chinese Medical Association in 2006.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Water swallow test> Level 3.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale-liquid | day 1 and day 42
  The Penetration-Aspiration Scale (PAS) was conducted under video fluoroscopic swallowing study. PAS is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The PAS scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.
  In this assessment, we used 60% barium sulfate suspension A higher level of PAS indicated a severer dysphagia.
Penetration-Aspiration Scale-paste | day 1 and day 42
  The Penetration-Aspiration Scale (PAS) was conducted under video fluoroscopic swallowing study. PAS is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The PAS scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.
  In this assessment, we used 180% barium sulfate suspension A higher level of PAS indicated a severer dysphagia.

SECONDARY OUTCOMES:
Swallowing time-The oral transit time-liquid | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The liquid (60% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-The oral transit time-paste | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The paste (180% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-swallowing reaction time-liquid | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The liquid (60% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-pharyngeal transit time -liquid | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The liquid (60% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-laryngeal closure duration-liquid | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The liquid (60% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-swallowing reaction time-paste | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The paste (180% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-pharyngeal transit time-paste | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The paste (180% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Swallowing time-laryngeal closure duration-paste | day 1 and day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The paste (180% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
Nutritional status-body mass index | day 1 and day 42
  Patients' body mass index was assessed with the physical check, with the combination of height and body weight. as kg/m^2, reference range: 18.5 kg/m2≤BMI<24 kg/m2.
  Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Nutritional status-Serum Albumin | day 1 and day 42
  Patients' Serum Albumin was assessed from the routine blood test, reference range: 35~50 g/L.Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Nutritional status-Prealbumin | day 1 and day 42
  Patients' Prealbumin was assessed from the routine blood test, reference range: 200~400 mg/L.Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Nutritional status-Hemoglobin | day 1 and day 42
  Patients' Hemoglobin was assessed from the routine blood test, reference range: males: 120~160 g/L, females: 110~150 g/L. Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Standardized Swallowing Assessment | day 1 and day 42
  The Standardized Swallowing Assessment (SSA) consists of three main parts: clinical examination, 5ml water swallow, and daily water intake assessment. The highest score is 46 points, the lowest is 18 points, with lower scores indicating better swallowing function.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Quanmi Hos., Pingdong, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng HJ, Zhao WJ, Luo PC, Zhang XY, Luo SY, Li Y, Li HP, Wang LG, Zeng X. Acupuncture Therapy on Dysphagia in Patients with Parkinson's Disease: A Randomized Controlled Study. Chin J Integr Med. 2025 Mar;31(3):261-269. doi: 10.1007/s11655-024-3668-x. Epub 2024 Sep 21. PMID 39305459